CLINICAL TRIAL: NCT05473039
Title: OvoVid Study: Effect of a Multivitamin Supplement With Probiotic (Seidivid Ferty4®) on Oocyte Retrieval and Quality in Oocyte Donors. Double-blind Randomized Placebo-controlled Clinical Trial
Brief Title: Effect of a Multivitamin Supplement With Probiotic (Seidivid Ferty4®) on Oocyte Retrieval and Quality
Acronym: OvoVid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEID S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OVOVID-FERTY4-2022-01
Record Dates: First submitted 2022-06-27; First posted 2022-07-25 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Reproductive Techniques, Assisted
Keywords: oocyte maduration; oocyte donation; dietary supplement
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, double-blind, placebo-controlled clinical trial with a dietary supplement with probiotics, with two parallel group of subjects.
  Based on previous studies, considering this study as a non-inferiority versus placebo study the calculated sample size of subjects is 210 (105 subject for each arm).
  Once the informed consent is signed, the patient will be assigned a patient code and will be given the treatment box (white and with no label) corresponding to her code. The patient will start taking the study treatment (multivitamin supplement with probiotics or placebo) immediately after inclusion. Throughout the COH period the patient will continue taking the study supplement and will undergo the regular ultrasound controls of the egg donation program for evolutive control of the number and growth of follicles, without interruption until the day of the GnRH-agonist trigger.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study multivitamin product with probiotics (Seidivid Ferty4®) and placebo will be supplied as capsules with an identical external appearance packaged in blisters in a white box with no label, marked only with the study code and patient code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seidivid Ferty4 (Experimental): Patients included in this group will be administered dietary supplement Seidivid Ferty4 (2 capsules per day, as a single dose) for at least 30 days prior to controlled ovarian hyperstimulation and until the day of the agonist trigger (GnRH a).
  Interventions: Dietary Supplement: Seidivid Ferty4
- Placebo (Placebo Comparator): Patients included in this group will be administered placebo (2 capsules per day, as a single dose) for at least 30 days prior to controlled ovarian hyperstimulation and until the day of the agonist trigger (GnRH-a).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Seidivid Ferty4 — The patient will start taking the study treatment (multivitamin supplement with probiotics) immediately after inclusion. Throughout the COH period of the protocol (usual mean duration: 11 days) the patient will continue taking the diatary supplement, without interruption until the day of the GnRH-agonist trigger.
  Arms: Seidivid Ferty4
Other: Placebo — The patient will start taking the study treatment (placebo) immediately after inclusion. Throughout the COH period of the protocol (usual mean duration: 11 days) the patient will continue taking the treatment (placebo), without interruption until the day of the GnRH-agonist trigger.
  Arms: Placebo

SUMMARY:
This study evaluates the effect of pretreatment with a multivitamin supplement with probiotics (Seidivid Ferty4®) on oocyte retrieval in normo-responder patients undergoing controlled ovarian hyperstimulation (COH) for oocyte donation, considering both the total number of oocytes retrieved and the number of mature oocytes retrieved, that is, in metaphase II (MII).

DETAILED DESCRIPTION:
Patients will be recruited on the day they are going to start the egg donation program. The patient will start taking the study treatment (multivitamin supplement with probiotics or placebo) immediately after inclusion and will call the site to initiate the oocyte donation protocol approximately 30 days after enrollment. Throughout the COH period of the protocol the patient will continue taking the study supplement (or placebo), without interruption until the day of the GnRH-agonist trigger. The administration of the agonist will be as a single dose, 36 hours before follicular puncture for the retrieval of mature eggs. Then, the retrieved oocytes will be denuded and examined by light microscopy to assess their quality. The evaluation will carried out by two different embryologists, blinded to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing COH for egg donation cycles
* Signing of Informed Consent
* Age 18-34 years
* Body mass index between 18-29.9 kg/m2
* Meet the criteria for inclusion in the oocyte donation program of the Next Fertility center
* Ultrasound antral follicle count before COH of ≥15 follicles

Exclusion Criteria:

* Patients excluded from the oocyte donation program
* Untreated sexually transmitted disease, HIV, HCV, HBV positive serology
* Blood disorders, neurodegenerative/psychiatric diseases, fragile X syndrome, oncological diseases, endometriosis.
* Polycystic ovary syndrome
* Oligomenorrhea (<1 menstrual cycle in 3 months)
* Diabetic patients

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Quintero, Ph, Study Director — NextFertility Valencia
Locations (1):
- NextFertility, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available because the voluntary participating oocyte donors are healthy women and are not amenable to further follow-up.

REFERENCES:
- [Derived] Bonta S, Maggi S, Rodriguez R, Jimenez R, Villaquiran AM, Pla E, Fuentes R, Luque MD, Ferrer J, Quintero L. Ovovid trial: the effect of a probiotic micronutrients supplement on oocyte retrieval and quality in oocyte donors. A double blind, randomized controlled trial. J Assist Reprod Genet. 2025 Dec 9. doi: 10.1007/s10815-025-03763-4. Online ahead of print. PMID 41361728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Seidivid Ferty4 | Placebo
Started | 98 | 98
Completed | 70 | 65
Not Completed | 28 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seidivid Ferty4 | Placebo | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data not available for 1 patient in placebo group
  years
    number analyzed (Participants) | 98 | 97 | 195
    (all) | 24.06 (4.09) | 23.10 (3.24) | 23.58 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 98 | 196
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 98 | 98 | 196
Region of Enrollment [Number; unit: participants]
  Spain | 98 | 98 | 196
Baseline Fasting Glucose [Mean (Standard Deviation); unit: mg/dl] — Fasting blood glucose at the time of study inclusion Population: Data not available for 47 participants
  mg/dl
    number analyzed (Participants) | 80 | 69 | 149
    (all) | 81.21 (8.48) | 79.91 (9.27) | 80.61 (8.85)
Number of Antral Follicles at Study Inclusion [Mean (Standard Deviation); unit: antral follicles] — Ultrasound antral follicle count at study inclusión Population: Data not available for 2 participants
  antral follicles
    number analyzed (Participants) | 98 | 96 | 194
    (all) | 22.30 (4.73) | 21.33 (4.54) | 21.82 (4.65)
Baseline AST [Mean (Standard Deviation); unit: U/L] — Serum aspartate aminotransferase (AST) levels at the time of study inclusión Population: Data not available for 18 participants
  U/L
    number analyzed (Participants) | 90 | 88 | 178
    (all) | 21.31 (13.78) | 19.88 (6.42) | 20.60 (10.78)
Baseline ALT [Mean (Standard Deviation); unit: U/L] — Serum alanine aminotransferase (ALT) levels at the time of study inclusión Population: Data not available for 18 participants
  U/L
    number analyzed (Participants) | 90 | 88 | 178
    (all) | 17.72 (10.07) | 16.80 (8.26) | 17.26 (9.20)
Baseline Cholesterol LDL [Mean (Standard Deviation); unit: mg/dl] — Cholesterol LDL at the time of study inclusión Population: Data not available for 18 participants
  mg/dl
    number analyzed (Participants) | 90 | 88 | 178
    (all) | 89.32 (21.48) | 87.83 (23.25) | 88.58 (22.32)
Baseline Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Total cholesterol at the time of study inclusión Population: Data not available for 18 participants
  mg/dL
    number analyzed (Participants) | 90 | 88 | 178
    (all) | 165.91 (29.74) | 164.40 (31.29) | 165.16 (29.74)

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Description: Total number of oocytes retrieved in the follicular puncture
Time Frame: Through study completion, an average of 42 days
Population: Only patients who completed the study and underwent follicular puncture
Measure: Geometric Mean (Standard Deviation); unit: oocytes retrieved
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 70 | 65
oocytes retrieved | 24.77 (10.96) | 22.57 (9.12)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.2629, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Mature (MII) Oocytes Retrieved
Description: Total number of mature oocytes (metaphase II, or MII) retrieved in the follicular puncture
Time Frame: Through study completion, an average of 42 days
Population: Only patients who completed the study and underwent follicular puncture
Measure: Geometric Mean (Standard Deviation); unit: mature oocytes
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 70 | 65
mature oocytes | 20.41 (9.32) | 18.86 (8.47)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.3582, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Good Quality Oocytes
Description: Number of oocytes MII without dimorphisms
Time Frame: Through study completion, an average of 42 days
Population: Only patients who completed the study underwent follicular puncture and retrieved MII oocytes. One case was excluded because no mature oocytes were retrieved.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 69 | 65
oocytes | 17.00 (7.67) | 15.43 (8.20)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.2187, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Oocytes With Dimorphisms
Description: Number of mature oocytes MII with dimorphisms
Time Frame: Through study completion, an average of 42 days
Population: Only patients who completed the study and underwent follicular puncture, and who specified whether the oocytes had dysmorphisms. One case was excluded because no mature oocytes were obtained, and three cases were excluded because the number of dysmorphic oocytes was not specified.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 68 | 63
oocytes | 3.71 (4.41) | 3.46 (4.66)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.3005, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Follicles at the Time of Trigger Administration
Description: Ultrasound follicle count at the time of trigger administration
Time Frame: Through trigger administration, an average of 40 days
Measure: Mean (Standard Deviation); unit: follicle count
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 75 | 65
follicle count | 28.01 (10.41) | 24.8 (7.08)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.0314, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Fasting Glucose After 30 Days of Treatment With Dietary Supplement.
Description: Fasting blood glucose at the start of controlled ovarian hyperstimulation (COH)
Time Frame: Through COH start, an average of 30 days
Population: Only patients with fasting glucose data recorded at baseline and at 30 days were analysed.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 69 | 61
mg/dl | 81.49 (13.04) | 82.48 (9.02)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.9214, t-test, 2 sided
Statistical Analysis 2: Comparison: Seidivid Ferty4; Fasting glucose at the start of COH compared to baseline fasting glucose; Test type: Superiority; p = 0.042, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Fasting glucose at the start of COH compared to baseline fasting glucose; Test type: Superiority; p < 0.001, t-test, 2 sided

7. Secondary Outcome: AST After 30 Days of Treatment With Dietary Supplement.
Description: Serum aspartate aminotransferase (AST) levels at the time of controlled ovarian hyperstimulation (COH) start
Time Frame: Through COH start, an average of 30 days
Population: Only patients with AST data recorded at baseline and at 30 days were analysed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 77 | 76
U/L | 20.38 (5.79) | 20.37 (6.14)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.59695, t-test, 2 sided
Statistical Analysis 2: Comparison: Seidivid Ferty4; AST at the start of COH compared to baseline AST; Test type: Superiority; p = 0.466503, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; AST at the start of COH compared to baseline AST; Test type: Superiority; p = 0.959877, t-test, 2 sided

8. Secondary Outcome: ALT After 30 Days of Treatment With Dietary Supplement.
Description: Serum alanine aminotransferase (ALT) levels at the time of controlled ovarian hyperstimulation (COH) start
Time Frame: Through COH start, an average of 30 days
Population: Only patients with ALT data recorded at baseline and at 30 days were analysed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 77 | 75
U/L | 19.14 (8.75) | 16.84 (6.13)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.062810, t-test, 2 sided
Statistical Analysis 2: Comparison: Seidivid Ferty4; ALT at the start of COH compared to baseline ALT; Test type: Superiority; p = 0.417757, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; ALT at the start of COH compared to baseline ALT; Test type: Superiority; p = 0.968525, t-test, 2 sided

9. Secondary Outcome: Cholesterol After 30 Days of Treatment With Dietary Supplement.
Description: Total cholesterol at the time of controlled ovarian hyperstimulation (COH) start
Time Frame: Through COH start, an average of 30 days
Population: Only patients with total cholesterol data recorded at baseline and at 30 days were analysed.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 76 | 76
mg/dl | 167.89 (29.66) | 170.17 (31.33)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.686488, t-test, 2 sided
Statistical Analysis 2: Comparison: Seidivid Ferty4; Cholesterol at the start of COH compared to baseline cholesterol; Test type: Superiority; p = 0.395120, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Cholesterol at the start of COH compared to baseline cholesterol; Test type: Superiority; p = 0.127135, t-test, 2 sided

10. Secondary Outcome: LH at the Time of COH Start
Description: Plasma levels of luteinizing hormone (LH) at the time of controlled ovarian hyperstimulation (COH) start
Time Frame: Through COH start, an average of 30 days
Measure: Mean (Standard Deviation); unit: mUI/ml
Arm/Group | Seidivid Ferty4 | Placebo
Number analyzed (Participants) | 77 | 75
mUI/ml | 6.55 (4.16) | 5.69 (3.96)
Statistical Analysis 1: Comparison: Seidivid Ferty4 vs Placebo; Test type: Superiority; p = 0.257496, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 42 days
Description: Adverse events described by patients and recorded by the investigator at each control visit
Arm/Group | Seidivid Ferty4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 2/98 | 0/98
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seidivid Ferty4 (N=98) | Placebo (N=98)
Sleepiness (Nervous system disorders) | 1 (1) | 0 (0) — Mild sleepiness since the start of treatment. Causal relationship to treatment: possible
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 — Mild skin eruptions appearing after 20 days of treatment. Relationship to treatment: possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT05473039/Prot_SAP_000.pdf